CLINICAL TRIAL: NCT01024231
Title: A Phase 1b, Open-label, Multicenter, Multidose, Dose-escalation Study of BMS-936558 (MDX-1106) in Combination With Ipilimumab in Subjects With Unresectable Stage III or Stage IV Malignant Melanoma
Brief Title: Dose-escalation Study of Combination BMS-936558 (MDX-1106) and Ipilimumab in Subjects With Unresectable Stage III or Stage IV Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry); Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-004; (MDX1106-04) (Other: Medarex)
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: BMS-936558 (0.3 mg/kg)+Ipilimumab (3 mg/kg) (Experimental): BMS-936558 (MDX1106-04) 0.3 mg/kg solution, 60 minutes intravenous infusion every 3 (q3) weeks for 21 weeks in induction and every 12 (q12) weeks for 84 weeks in maintenance
  Ipilimumab (BMS-734016) 3 mg/kg solution, 90 minutes intravenous infusion q3 weeks for 9 weeks in induction and q12 weeks for 84 weeks in maintenance
  Interventions: Drug: BMS-936558 (MDX1106-04); Drug: Ipilimumab
- Cohort 2: BMS-936558 (1 mg/kg)+Ipilimumab (3 mg/kg) (Experimental): Ipilimumab (BMS-734016) 3 mg/kg solution, 90 minutes intravenous infusion, q3 weeks for 9 weeks in induction and q12 weeks for 84 weeks in maintenance
  BMS-936558 (MDX1106-04) 1 mg/kg solution, 60 minutes intravenous infusion, q3 weeks for 21 weeks in induction and q12 weeks for 84 weeks in maintenance
  Interventions: Drug: BMS-936558 (MDX1106-04); Drug: Ipilimumab
- Cohort 3: BMS-936558 (3 mg/kg)+Ipilimumab (3 mg/kg) (Experimental): Ipilimumab (BMS-734016) 3 mg/kg solution, 90 minutes intravenous infusion, q3 weeks for 9 weeks in induction and q12 weeks for 84 weeks in maintenance
  BMS-936558 (MDX1106-04) 3 mg/kg solution, 60 minutes intravenous infusion, q3 weeks for 21 weeks in induction and q12 weeks for 84 weeks in maintenance
  Interventions: Drug: BMS-936558 (MDX1106-04); Drug: Ipilimumab
- Cohort 4: BMS-936558 (10 mg/kg)+Ipilimumab (3 mg/kg) (Experimental): BMS-936558 (MDX1106-04) 10 mg/kg solution, 60 minutes intravenous infusion, q3 weeks for 21 weeks in induction and q12 weeks for 84 weeks in maintenance
  Ipilimumab (BMS-734016) 3 mg/kg solution, 90 minutes intravenous infusion, q3 weeks for 9 weeks in induction and q12 weeks for 84 weeks in maintenance
  Interventions: Drug: BMS-936558 (MDX1106-04); Drug: Ipilimumab
- Cohort 5: BMS-936558 (10 mg/kg)+Ipilimumab (10 mg/kg) (Experimental): BMS-936558 (MDX1106-04) 10 mg/kg solution, 60 minutes intravenous infusion, q3 weeks for 21 weeks in induction and q12 weeks for 84 weeks in maintenance
  Ipilimumab (BMS-734016) 10 mg/kg solution, 90 minutes intravenous infusion, q3 weeks for 9 weeks in induction and q12 weeks for 84 weeks in maintenance
  Interventions: Drug: BMS-936558 (MDX1106-04); Drug: Ipilimumab
- Cohort 6: BMS-936558 (1 mg/kg) (Experimental): BMS-936558 (MDX1106-04) 1 mg/kg solution, 60 minutes intravenous infusion, once q2 weeks for a total maximal duration of 96 weeks
  Interventions: Drug: BMS-936558 (MDX1106-04)
- Cohort 7: BMS-936558 (3 mg/kg) (Experimental): BMS-936558 (MDX1106-04) 3 mg/kg solution, 60 minutes intravenous infusion, once q2 weeks for a total maximal duration of 96 weeks
  Interventions: Drug: BMS-936558 (MDX1106-04)
- Cohort 8: Nivolumab+Ipilimumab (Experimental): Nivolumab 1 mg/kg and Ipilimumab 3 mg/kg solution intravenously q3 weeks, 4 doses for 12 weeks
  Followed by Nivolumab 3 mg/kg solution alone intravenously q2 weeks, 48 doses for a maximum of 96 weeks
  Interventions: Drug: BMS-936558 (MDX1106-04); Drug: Ipilimumab

INTERVENTIONS:
Drug: BMS-936558 (MDX1106-04)
  Other Names: Nivolumab
Drug: Ipilimumab
  Other Names: BMS-734016
  Arms: Cohort 1: BMS-936558 (0.3 mg/kg)+Ipilimumab (3 mg/kg); Cohort 2: BMS-936558 (1 mg/kg)+Ipilimumab (3 mg/kg); Cohort 3: BMS-936558 (3 mg/kg)+Ipilimumab (3 mg/kg); Cohort 4: BMS-936558 (10 mg/kg)+Ipilimumab (3 mg/kg); Cohort 5: BMS-936558 (10 mg/kg)+Ipilimumab (10 mg/kg); Cohort 8: Nivolumab+Ipilimumab

SUMMARY:
The purpose of this study is to determine the safety and tolerability of treatment with BMS-936558 (MDX-1106) in combination with Ipilimumab (BMS-734016) when given at the same time or as a sequenced regimen in subjects with unresectable Stage III or Stage IV malignant melanoma (MEL)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologic diagnosis of malignant melanoma (MEL)
* Measurable unresectable Stage III or IV MEL
* ECOG performance status score of 0 or 1
* Life expectancy ≥4 months
* For those enrolled in amendment 5 and later, tumor tissue (archival or recent acquisition) must be available
* For Cohorts 1-5, subjects may have been treated with up to 3 prior systemic standard treatments for metastatic melanoma not including any post-incisional adjuvant therapy. Subjects may be treatment naïve. All metastatic melanoma regardless of primary site of disease will be allowed
* For Cohorts 6-7, subjects may have been treated with up to 3 prior systemic standard treatments for metastatic melanoma; this does not include any post-incisional adjuvant therapy. Specifically, subjects must have received ≥3 doses of Ipilimumab therapy and the last dose having been administered within 4-12 weeks of initiation of study treatment

Exclusion Criteria:

* History of severe hypersensitivity reactions to other mAbs
* Prior malignancy active within the previous 2 years except for localized cancers that are considered to have been cured and in the opinion of the investigator present a low risk for recurrence
* Active autoimmune disease or a history of known or suspected autoimmune disease
* History of recently active diverticulitis or symptomatic peptic ulcer disease and history of adrenal insufficiency
* Regular narcotic analgesia
* Active, untreated central nervous system metastasis
* For subjects enrolled in Cohorts 1-5, prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibody
* For subjects enrolled in Cohorts 6-7, prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CD137 antibodies
* Any non-oncology vaccine therapy used for prevention of infectious disease
* Concomitant therapy with any other anti-cancer therapy, concurrent medical conditions requiring use of immunosuppressive medications or use of other investigational drugs
* Positive tests for human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS), hepatitis B, hepatitis C
* Subjects weighing ≥125 kg are excluded from Cohort 5
* Subjects in Cohorts 6 and 7 must have received Ipilimumab monotherapy immediately prior to study entry, but must not have received that Ipilimumab as part of a clinical trial
* Subjects with ocular melanoma are excluded from Cohort 8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-12-14 (Actual); Primary Completion 2014-02-04 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Yale University School Of Medicine, New Haven, Connecticut
  - Medstar Georgetown-Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Memorial Sloan Kettering Nassau, New York, New York
  - Hillman Cancer Research Pavilion, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Long GV, Larkin J, Schadendorf D, Grob JJ, Lao CD, Marquez-Rodas I, Wagstaff J, Lebbe C, Pigozzo J, Robert C, Ascierto PA, Atkinson V, Postow MA, Atkins MB, Sznol M, Callahan MK, Topalian SL, Sosman JA, Kotapati S, Thakkar PK, Ritchings C, Pe Benito M, Re S, Soleymani S, Hodi FS. Pooled Long-Term Outcomes With Nivolumab Plus Ipilimumab or Nivolumab Alone in Patients With Advanced Melanoma. J Clin Oncol. 2025 Mar 10;43(8):938-948. doi: 10.1200/JCO.24.00400. Epub 2024 Nov 6. PMID 39504507
- [Derived] Callahan MK, Kluger H, Postow MA, Segal NH, Lesokhin A, Atkins MB, Kirkwood JM, Krishnan S, Bhore R, Horak C, Wolchok JD, Sznol M. Nivolumab Plus Ipilimumab in Patients With Advanced Melanoma: Updated Survival, Response, and Safety Data in a Phase I Dose-Escalation Study. J Clin Oncol. 2018 Feb 1;36(4):391-398. doi: 10.1200/JCO.2017.72.2850. Epub 2017 Oct 17. PMID 29040030
- [Derived] Nguyen AT, Elia M, Materin MA, Sznol M, Chow J. Cyclosporine for Dry Eye Associated With Nivolumab: A Case Progressing to Corneal Perforation. Cornea. 2016 Mar;35(3):399-401. doi: 10.1097/ICO.0000000000000724. PMID 26771550
- [Derived] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 127 Randomized and Treated
Groups:
- Cohort 1: 0.3 mg/kg of BMS-936558 (MDX-1106) + 3 mg/kg of ipilimumab
- Cohort 2: 1 mg/kg of BMS-936558 (MDX-1106) + 3 mg/kg of ipilimumab
- Cohort 2a: 3 mg/kg of BMS-936558 (MDX-1106) + 1 mg/kg of ipilimumab
- Cohort 3: 3 mg/kg of BMS-936558 (MDX-1106) + 3 mg/kg of ipilimumab
- Cohort 6: 1mg/kg of BMS-936558 (MDX-1106)
- Cohorot 7: 3 mg/kg of BMS-936558 (MDX-1106)
- Cohort 8: 1 mg/kg of BMS-936558 (MDX-1106) in combination with 3 mg/kg of ipilimumab every 3 weeks for 4 doses
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohorot 7 | Cohort 8
Started | 14 | 17 | 16 | 6 | 17 | 16 | 41
Completed | 2 | 2 | 6 | 1 | 0 | 0 | 20
Not Completed | 12 | 15 | 10 | 5 | 17 | 16 | 21
Not completed — Other Reasons | 1 | 2 | 0 | 0 | 2 | 0 | 1
Not completed — Maximum Clinical Benefit | 1 | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Disease Progression | 3 | 1 | 3 | 0 | 4 | 11 | 6
Not completed — AE unrelated to Study Drug | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — No longer meets criteria | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Study Drug Toxicity | 1 | 6 | 6 | 4 | 2 | 0 | 7
Not completed — Death | 6 | 2 | 1 | 0 | 4 | 3 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrew Consent | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Continuing on Treatment | 0 | 0 | 0 | 0 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohorot 7 | Cohort 8 | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 17 | 16 | 41 | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (9.58) | 53.5 (14.14) | 59.1 (14.65) | 56.2 (11.99) | 63.9 (14.37) | 60.6 (17.56) | 55.2 (15.83) | 57.6 (13.78)
Age, Customized [Count of Participants; unit: Participants]
  <65 Years | 11 | 14 | 10 | 5 | 7 | 11 | 32 | 90
  ≥ 65 Years | 3 | 3 | 6 | 1 | 10 | 5 | 9 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 4 | 5 | 8 | 7 | 23 | 59
  Male | 9 | 10 | 12 | 1 | 9 | 9 | 18 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 14 | 17 | 16 | 6 | 15 | 16 | 39 | 123
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 14 | 17 | 16 | 6 | 16 | 16 | 37 | 122
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: incidence of all cause and treatment related adverse events
Time Frame: Up to 3 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Groups:
- Any BMS and Ipi Combo: All participants who received treatment in Cohorts 1 through 3
- Only BMS: combined total of participants who receive BMS only
- Any BMS/Ipi: All participants who received both BMS and Ipi
- Total: All Participants who received treatment in any cohort combined
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Participants
  All Cause | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
  Treatment Related | 13 | 17 | 15 | 6 | 51 | 15 | 13 | 28 | 40 | 91 | 119

2. Primary Outcome: Number of Participants With a Serious Adverse Event (AE)
Description: incidence of all cause and treatment related serious adverse events
Time Frame: Up to 3 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Participants
  All Cause | 10 | 15 | 10 | 5 | 40 | 9 | 10 | 19 | 26 | 66 | 85
  Treatment Related | 5 | 13 | 9 | 4 | 31 | 4 | 4 | 8 | 18 | 49 | 57

3. Primary Outcome: Number of Participants With an Adverse Event (AE) Which Lead to Discontinuation
Description: incidence of all cause and treatment related adverse events which lead to discontinuation
Time Frame: Up to 3 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Participants
  All Cause | 2 | 8 | 5 | 1 | 16 | 5 | 1 | 6 | 13 | 29 | 35
  Treatment Related | 2 | 6 | 5 | 1 | 14 | 2 | 0 | 2 | 11 | 25 | 27

4. Primary Outcome: Number of Deaths
Description: incidence of all cause and treatment related deaths
Time Frame: Up to 3 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Participants
  All Cause | 8 | 4 | 2 | 0 | 14 | 7 | 8 | 15 | 8 | 22 | 37
  Treatment Related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

5. Primary Outcome: Number of Participants With Select AEs
Description: incidence of all cause and treatment related Adverse events in certain organ systems
Time Frame: Up to 3 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Participants
  Endrocrine | 2 | 5 | 3 | 3 | 13 | 4 | 1 | 5 | 12 | 25 | 30
  Gastrointestinal | 5 | 7 | 10 | 4 | 26 | 3 | 4 | 7 | 20 | 46 | 53
  Hepatic | 5 | 6 | 4 | 3 | 18 | 1 | 1 | 2 | 8 | 26 | 28
  Pulmonary | 1 | 2 | 1 | 0 | 4 | 0 | 1 | 1 | 2 | 6 | 7
  Renal | 2 | 1 | 1 | 1 | 5 | 0 | 1 | 1 | 1 | 6 | 7
  Skin | 12 | 15 | 15 | 4 | 46 | 8 | 10 | 18 | 34 | 80 | 98
  Hypersensitivity/Infusion Reaction | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 3 | 5

6. Primary Outcome: Laboratory Abnormalities: Specific Liver Tests
Description: Number of Participants with On-Treatment Laboratory Abnormalities in Specific Liver Tests Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Upper Limit of Normal (ULN)
Time Frame: Up to 3 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Participants
  ALT or AST > 3xULN | 1 | 0 | 2 | 3 | 6 | 0 | 1 | 1 | 6 | 12 | 13
  ALT or AST > 5xULN | 3 | 1 | 1 | 1 | 6 | 0 | 0 | 0 | 5 | 11 | 11
  ALT or AST > 10xULN | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 5 | 5
  ALT or AST > 20xULN | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4 | 4
  Total Bilirubin (Tbili) > 2xULN | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 3
  ALT or AST > 3xULN w/ Tbili > 2xULN within 1 day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

7. Primary Outcome: Laboratory Abnormalities: Specific Thyroid Tests
Description: Number of Participants with On-Treatment Laboratory Abnormalities in Specific Thyroid Tests Free T3 (FT3) Free T4 (FT4) Lower Limit of Normal (LLN)
Time Frame: Up to 3 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Participants
  TSH > ULN | 7 | 9 | 7 | 3 | 26 | 4 | 3 | 7 | 8 | 34 | 41
  TSH > ULN with TSH≤ ULN @ Baseline | 3 | 6 | 7 | 1 | 17 | 3 | 1 | 4 | 6 | 23 | 27
  TSH > ULN: WITH ALL OTHER T3/T4 TEST ≥ LLN | 7 | 9 | 7 | 2 | 25 | 4 | 3 | 7 | 8 | 33 | 40
  TSH > ULN: WITH AT LEAST ONE T3/T4 TEST < LLN | 5 | 6 | 5 | 2 | 18 | 2 | 1 | 3 | 5 | 23 | 26
  TSH > ULN: WITH FT3/FT4 TEST MISSING | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TSH < LLN | 3 | 7 | 7 | 3 | 20 | 4 | 1 | 5 | 14 | 34 | 39
  TSH < LLN: WITH TSH >= LLN AT BASELINE | 3 | 7 | 7 | 3 | 20 | 3 | 0 | 3 | 14 | 34 | 37
  TSH < LLN: WITH ALL OTHER FT3/FT4 TEST ≤ ULN | 2 | 6 | 6 | 3 | 17 | 4 | 1 | 5 | 11 | 28 | 33
  TSH < LLN: WITH AT LEAST ONE T3/T4 TEST > ULN | 3 | 3 | 3 | 2 | 11 | 2 | 0 | 2 | 8 | 19 | 21
  TSH < LLN: WITH FT3/FT4 TEST MISSING | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Objective Response Rate
Description: the total number of participants whose best overall response (BOR) is either irCR or irPR divided by the total number of response-evaluable participants.
Time Frame: Up to 3 years
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Percentage of Participants | 21 [4.7 to 50.8] | 47 [23.0 to 72.2] | 50 [24.7 to 75.3] | 50 [11.8 to 88.2] | 42 [28.1 to 55.9] | 53 [27.8 to 77.0] | 19 [4.0 to 45.6] | 36 [20.4 to 54.9] | 44 [28.5 to 60.3] | 43 [32.4 to 53.2] | 41 [32.3 to 50.0]

9. Secondary Outcome: Time to Response
Description: the time from the first dose of study drug until the first documentation of irCR or irPR, as related to current database lock date or most current tumor measurement
Time Frame: Up to 3 Years
Population: All Treated Participants
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 16 | 33 | 41 | 94 | 127
Weeks | 11.9 [11.9 to 12.9] | 11.9 [7.7 to 14.7] | 11.9 [7.0 to 18.7] | 12.3 [10.4 to 18.0] | 11.9 [7.0 to 18.7] | 8 [7.4 to 34.1] | 15.7 [7.7 to 16.0] | 9.6 [7.4 to 34.1] | 12.1 [11.0 to 24.1] | 12 [7.0 to 24.1] | 12 [7.0 to 34.1]

10. Secondary Outcome: Duration of Response
Description: the time from the first documented response (irCR or irPR) until progression or death, whichever occurs first. For participants who did not progress or die, duration of response will be censored on the date of the last tumor assessment.
Time Frame: from the first documented response (irCR or irPR) until progression or death
Population: All Treated Participants with a response
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 53 | 17 | 3 | 33 | 41 | 94 | 127
Weeks | NA [78.4 to NA] — Not a sufficient amount of responders to calculate median duration of response. | 105 [105 to 141] | 66.3 [66.3 to NA] — insufficient number of responders in order to derive 95%CI | 59.1 [31.3 to 86.9] | 105 [86.9 to 141] | 73.1 [73.1 to NA] — upper limit number not reached | 64.3 [NA to NA] — upper limit number not reached lower limit number: insufficient number of responders in order to derive 95%CI | 73.1 [64.3 to NA] — insufficient number of responders in order to derive 95%CI | NA [NA to NA] — Not a sufficient amount of responders to calculate median duration of response. lower limit number: insufficient number of responders in order to derive 95%CI | 105 [78.4 to 141] | 105 [78.4 to 141]

11. Secondary Outcome: Progression Free Survival
Description: the time from the first dose to the first observation of disease progression or death due to any cause. If a participant has not progressed or died at the time of analysis, PFS will be censored on the date of the last disease assessment. Participants who did not have any on-study tumor assessments and did not die will be censored on the date of the first dose of study medication.
Time Frame: 156 weeks
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 0 | 17 | 16 | 0 | 41 | 0
Weeks | 12.50 [11.60 to 47.90] | 64.40 [12.00 to 149.00] | 58.40 [12.00 to NA] — Upper limit number not reached | 33.55 [11.60 to 97.10] |  | 24.60 [8.10 to NA] — Upper limit number not reached | 12.15 [7.70 to 23.90] |  | 37.10 [12.90 to NA] — Upper limit number not reached |

12. Secondary Outcome: Number of Participants With an Anti-Drug Antibody (ADA) Response for Nivolumab (Nivo) and Ipilimumab (Ipi)
Description: Serum samples will be collected to evaluate the development of antibodies to BMS-936558 and to ipilimumab.
Time Frame: Up to 3 years
Population: All Treated Participants with baseline and at least one post baseline assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 13 | 17 | 16 | 5 | 51 | 15 | 12 | 27 | 35 | 86 | 113
Participants
  Baseline ADA Positive (nivo) | 1 | 1 | 2 | 0 | 4 | 1 | 0 | 1 | 1 | 5 | 6
  Baseline ADA Positive (ipi): number analyzed (Participants) | 13 | 17 | 16 | 5 | 51 | 14 | 11 | 25 | 32 | 83 | 108
  Baseline ADA Positive (ipi) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 3 | 3
  ADA Positive (nivo) | 6 | 10 | 4 | 0 | 20 | 4 | 1 | 5 | 10 | 30 | 35
  ADA Positive (ipi): number analyzed (Participants) | 13 | 17 | 16 | 5 | 51 | 14 | 11 | 25 | 32 | 83 | 108
  ADA Positive (ipi) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 4
  ADA Negative (nivo) | 7 | 7 | 12 | 5 | 31 | 11 | 11 | 22 | 25 | 56 | 78
  ADA Negative (ipi): number analyzed (Participants) | 13 | 17 | 16 | 5 | 51 | 14 | 11 | 25 | 32 | 83 | 108
  ADA Negative (ipi) | 12 | 17 | 16 | 5 | 50 | 13 | 10 | 23 | 31 | 81 | 104

13. Secondary Outcome: Peak and Trough Concentrations
Description: The peak and trough concentrations of BMS-936558 (MDX-1106) and ipilimumab in participants with quantifiable data
Time Frame: Up to 64 Weeks
Population: All Treated Participants with quantifiable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Any BMS and Ipi Combo | Cohort 6 | Cohorot 7 | Only BMS | Cohort 8 | Any BMS/Ipi | Total
Number analyzed (Participants) | 14 | 17 | 16 | 6 | 0 | 7 | 10 | 0 | 40 | 0 | 0
ug/mL
  Nivo Peak (Cmax): number analyzed (Participants) | 13 | 17 | 15 | 6 | 0 | 7 | 10 | 0 | 40 | 0 | 0
  Nivo Peak (Cmax) | 6.5 (17.2) | 21.5 (17.9) | 49.8 (24.7) | 63.4 (18.0) |  | 20.5 (64.5) | 97.7 (52.5) |  | 18.1 (38.1) |  |
  Nivo Trough (Cmin): number analyzed (Participants) | 5 | 11 | 9 | 3 | 0 | 6 | 10 | 0 | 13 | 0 | 0
  Nivo Trough (Cmin) | 1.5 (44.9) | 2.6 (94.4) | 27.7 (23.9) | 23.9 (37.5) |  | 13.2 (40.9) | 53.1 (49.8) |  | 5.9 (49.3) |  |
  Ipi Peak (Cmax): number analyzed (Participants) | 13 | 17 | 16 | 6 | 0 | 0 | 0 | 0 | 36 | 0 | 0
  Ipi Peak (Cmax) | 63.9 (17.7) | 68.5 (20.4) | 19.8 (40.6) | 63.2 (24.2) |  |  |  |  | 63.5 (31.5) |  |
  Ipi Trough (Cmin): number analyzed (Participants) | 14 | 14 | 15 | 4 | 0 | 0 | 0 | 0 | 33 | 0 | 0
  Ipi Trough (Cmin) | 9.7 (33.7) | 11.9 (29.5) | 3.6 (30.4) | 9.2 (34.4) |  |  |  |  | 9.8 (43.7) |  |

ADVERSE EVENTS:
Time Frame: Within 100 days of discontinuation of dosing or within 30 days of the last visit for screen failures (Approximately 3 years)
Description: The Following arms: Any BMS and Ipi Combo, Only BMS and Total, were left out of the AE section because the participants in those arms are reflected in the other arms.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohorot 7 | Cohort 8
All-Cause Mortality (participants affected / at risk) | 8/14 | 4/17 | 2/16 | 0/6 | 7/17 | 8/16 | 8/41
Serious Adverse Events (participants affected / at risk) | 10/14 | 15/17 | 10/16 | 5/6 | 9/17 | 10/16 | 26/41
Other Adverse Events (participants affected / at risk) | 14/14 | 17/17 | 16/16 | 6/6 | 17/17 | 15/16 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=14) | Cohort 2 (N=17) | Cohort 2a (N=16) | Cohort 3 (N=6) | Cohort 6 (N=17) | Cohorot 7 (N=16) | Cohort 8 (N=41)
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0 | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease Progression (General disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 2
Pyrexia (General disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 2
Alanine Aminotransferase Increased (Investigations) | 3 | 3 | 2 | 1 | 0 | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 3 | 3 | 2 | 1 | 0 | 0 | 2
Blood Creatinine Increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1
Superinfection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infections (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune Disorder (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Convulsions (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2
Appendix Disorders (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Amylase Increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 2 | 0
Lipase Increased (Investigations) | 0 | 1 | 2 | 1 | 1 | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2
Central Nervous System Necrosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chorioretinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Urea Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin 1 Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cerebral Ischemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 0 | 0 | 7
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Sudden Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone Lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cognitive Disorders (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hospitalizations (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiorgan Failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Edema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterococcal Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastasis to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Central Nervous System Hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=14) | Cohort 2 (N=17) | Cohort 2a (N=16) | Cohort 3 (N=6) | Cohort 6 (N=17) | Cohorot 7 (N=16) | Cohort 8 (N=41)
Nausea (Gastrointestinal disorders) | 7 | 5 | 4 | 3 | 4 | 6 | 20
Diarrhea (Gastrointestinal disorders) | 5 | 6 | 8 | 4 | 3 | 4 | 17
Constipation (Gastrointestinal disorders) | 4 | 4 | 4 | 2 | 2 | 4 | 10
Abdominal Pain (Gastrointestinal disorders) | 3 | 3 | 3 | 1 | 0 | 1 | 11
Vomiting (Gastrointestinal disorders) | 3 | 3 | 3 | 1 | 0 | 1 | 10
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 2 | 2 | 6
Flatulence (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 6
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tongue Ulceration (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Anal Pruritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip Dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue Discoloration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue Edema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 11 | 11 | 4 | 7 | 5 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 11 | 12 | 3 | 4 | 4 | 22
Vitiligo (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 1 | 0 | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 3 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 5
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Butterfly Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hair Color Changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lichenoid Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 9 | 11 | 7 | 4 | 9 | 7 | 26
Pyrexia (General disorders) | 5 | 7 | 3 | 4 | 2 | 4 | 14
Chills (General disorders) | 3 | 5 | 1 | 0 | 1 | 2 | 7
Edema Peripheral (General disorders) | 2 | 2 | 1 | 1 | 1 | 3 | 4
Pain (General disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 2
Asthenia (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 2
Edema (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 2
Chest Pain (General disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Chest Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Influenza Like Illness (General disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Xerosis (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Axillary Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Local Swelling (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Catheter Site Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early Satiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling Jittery (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sensation of Foreign Body (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 7 | 2 | 5 | 6 | 17
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 1 | 1 | 2 | 7
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 6
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1 | 0 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 4
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthalgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3 | 2 | 4 | 7 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 2 | 2 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 3 | 3 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 2 | 0 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 0 | 0 | 1 | 4
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase Increased (Investigations) | 2 | 4 | 3 | 4 | 2 | 1 | 8
Amylase Increased (Investigations) | 2 | 4 | 2 | 3 | 1 | 0 | 6
Aspartate Aminotransferase Increased (Investigations) | 2 | 1 | 1 | 4 | 1 | 0 | 7
Weight Decreased (Investigations) | 2 | 1 | 3 | 2 | 1 | 2 | 5
Alanine Aminotransferase Increased (Investigations) | 1 | 4 | 0 | 2 | 0 | 1 | 7
Hemoglobin Decreased (Investigations) | 1 | 1 | 0 | 1 | 1 | 1 | 3
Weight Increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1 | 3
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 6
Blood Alkaline Phosphatase Increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 3
Blood Creatinine Increased (Investigations) | 2 | 1 | 0 | 1 | 0 | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Electrocardiogram QT Prolonged (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
International Normalized Ratio Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood Albumin Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Phosphorus Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Potassium Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Testosterone Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Uric Acid Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breath Sounds Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest X-Ray Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal Test Positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid Function Test Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 8 | 4 | 4 | 1 | 3 | 13
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 0 | 2 | 3 | 4
Neuropathy Peripheral (Nervous system disorders) | 4 | 3 | 0 | 0 | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 3 | 2 | 0 | 0 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness Postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine with Aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mononeuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Narcolepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 4 | 3 | 0 | 2 | 1 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 2 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infections (Infections and infestations) | 1 | 2 | 1 | 1 | 2 | 1 | 3
Urinary Tract Infections (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Oral Herpes (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Herpes Zoster (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis Orbital (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia Bacteremia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 4
Dry Eye (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 1
Uveitis (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Ocular Hyperemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Eye Pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye Swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid Margin Crusting (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ophthalmoplegia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 6
Hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 3
Thyroiditis (Endocrine disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 3 | 0 | 0 | 2 | 2
Hypotension (Vascular disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Confusional State (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Mood Altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radiation Necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radiation Skin Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Micturition Urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urethral Discharge (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Tract Disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hearing Impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ear Pruritus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast Cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polymenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-08-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT01024231/SAP_000.pdf
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT01024231/Prot_001.pdf